CLINICAL TRIAL: NCT00740363
Title: The Effect of Sitagliptin Treatment on Glucose Metabolism and Endothelial Function in Renal Transplant Recipients - JANUVIA-08
Brief Title: Sitagliptin in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JANUVIA-08
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Glucose Intolerance
Keywords: renal transplantation; diabetes; glucose intolerance; impaired glucose tolerance
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients will receive 4 weeks of treatment with sitagliptin once daily
  Interventions: Drug: sitagliptin
- B (Placebo Comparator): No treatment for 4 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sitagliptin — Once daily sitagliptin. If GFR>50 ml/min/1.73m2: 100 mg/day. If GFR from 25 to 49 ml/min/1.3m2: 50 mg/day
  Other Names: Januvia
  Arms: A
Drug: placebo — No active sitagliptin treatment for 4 weeks
  Arms: B

SUMMARY:
The major cause of premature death in renal transplant recipients is cardiovascular disease. Sitagliptin stimulates insulin secretion and inhibits glucagon release, two central mechanisms in PTDM by interaction with a hormone system (incretins) that just recently it has become possible to modulate by drugs. Sitagliptin therefore is an interesting additional drug for the treatment of posttransplant diabetes mellitus in transplanted patients.

The primary objective of the present study is to investigate the effect of sitagliptin on insulin secretion in renal transplant recipients.

Secondary objectives are to study the effect on insulin sensitivity, fasting blood glucose, endothelial function, CsA/Tac blood concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipient more than 1 year posttransplant with stable renal function (less than 20% deviation in serum creatinine the last 2 months) and stable prednisolone dose for the last 3 months before inclusion.
* Patients in need of (additional) oral anti-diabetic treatment:

  * New onset diabetes patients with fasting plasma glucose 7-8 mmol/ l, and/or 2-hr plasma glucose 12-18 mmol/l after an oral glucose tolerance test (OGTT)
  * Patients already on oral hypoglycemic therapy, but with HbA1c 8-11%
* 18 years of age.
* Male patient, or female patient without childbearing potential (surgically sterilized or postmenopausal) or, if female of childbearing potential, is not lactating, has a negative pregnancy test at screening and is willing to utilize an effective method of contraception throughout the study period and for 90 Days following discontinuation of the Study Drugs.
* Signed informed consent.

Exclusion Criteria:

* Treatment with insulin
* Severe liver disease.
* Estimated GFR < 25 ml/min/1.73 m2.
* Skin disorders that may influence laser Doppler flowmetry investigations.
* Pregnant or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Insulin secretion | 4 weeks

SECONDARY OUTCOMES:
Insulin sensitivity | 4 weeks
Fasting blood glucose | 4 weeks
Endothelial function | 4 weeks
Cyclosporine/tacrolimus blood concentrations | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Trond Jenssen, MD, Professor, Principal Investigator — Rikshospitalet Medical Center
Locations (1):
- Rikshospitalet Medical Center, Oslo, Norway

REFERENCES:
- [Derived] Lo C, Toyama T, Oshima M, Jun M, Chin KL, Hawley CM, Zoungas S. Glucose-lowering agents for treating pre-existing and new-onset diabetes in kidney transplant recipients. Cochrane Database Syst Rev. 2020 Jul 30;8(8):CD009966. doi: 10.1002/14651858.CD009966.pub3. PMID 32803882